CLINICAL TRIAL: NCT06706362
Title: Assessing the Utility of Prophylactic Antibiotics at Time of Urethral Bulking Using Bulkamid
Brief Title: Assessing the Utility of Prophylactic Antibiotics at Time of Urethral Bulking Using Bulkamid (Bulkamid Study)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Susanne Taege, MD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024H0366
Record Dates: First submitted 2024-11-11; First posted 2024-11-26 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Stress Urinary Incontinence
Keywords: Bulkamid; Urinary tract infections; Bactrim; Macrobid; Urethral bulking
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Tract Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Nitrofurantoin

STUDY DESIGN:
Intervention Model Description: a double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants, providers, investigators or outcome assessors will know to which of these groups participants are assigned. In case of an emergency, however, the study doctor can get this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bactrim or Macrobid (single dose) (Active Comparator): Bactrim (800/160mg) or Macrobid (100 mg) depending on participants' allergies
  Interventions: Drug: Bactrim or Macrobid
- Placebo (Placebo Comparator): Identical appearing placebo for a single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bactrim or Macrobid — Participants will be assigned to Bactrim or Macrobid depending on participants' allergies
  Arms: Bactrim or Macrobid (single dose)
Drug: Placebo — Participants will be assigned to identical appearing placebo
  Arms: Placebo

SUMMARY:
The primary aim of this study is to assess the utility of prophylactic oral antibiotics at time of Bulkamid transurethral bulking to reduce the incidence of urinary tract infection (UTI) in the immediate postoperative period. The secondary aims of the study include assessing UTI rates and success rates if patients require temporary indwelling catheter versus intermittent self-catheterization (ISC).

DETAILED DESCRIPTION:
Specific Aim 1: To determine if receiving prophylactic oral antibiotics at time of urethral bulking reduces the risk of post-operative urinary tract infection (UTI).

Patients will be randomized and blinded into two arms: oral antibiotic versus placebo. Patients will receive either the placebo pill or oral antibiotic in the pre-operative holding area prior to their procedure. Oral antibiotics will include trimethoprim/sulfamethoxazole (Bactrim, first line) or nitrofurantoin (Macrobid, second line), determined by patient allergies.

Specific Aim 2: To assess if factors such as patient discharge with ISC/indwelling foley or number of Bulkamid injection sites is correlated to improvement in Stress urinary incontinence (SUI) at 6 weeks postoperatively and at one year postoperatively.

Patients will complete a brief survey preoperative, at 6 weeks postoperatively after their procedure, and at 1 year postoperatively after their procedure. The survey will consist of prior validated urogynecologic surveys including the Pelvic Floor Disability Index/Urinary Distress Inventory (PFDI/UDI- 6) and the MESA questionnaires as well as an extended VAS scale to evaluate global improvement.

Specific Aim 3: To discern if any patient characteristics are associated with higher patient satisfaction following the procedure.

ELIGIBILITY:
Inclusion Criteria

* Patients evaluated by a pelvic floor specialist (either urogynecologist or urologist) at The Ohio State University with plans to undergo urethral bulking with Bulkamid for stress urinary incontinence or mixed urinary incontinence (stress predominant).
* Negative testing for UTI in pre-operative work-up (including either negative urine culture or urine dip negative for infection).
* Office evaluation with evidence of SUI either with urodynamic studies (UDS) or positive cough stress test (CST).
* Post-void residual volume of 150 mL or less (measured by either catheterization or bladder scan)

Exclusion Criteria

* Contraindications to both oral antibiotics including antibiotic allergies or significant renal disease
* Patient undergoing additional pelvic organ prolapse procedures or other urologic procedures concomitantly
* Recurrent UTIs, defined as 3 or more UTIs within the past 12 months or 2 UTIs within the past 6 months
* Patients currently taking daily antibiotic prophylaxis for any reason
* Non-English speaking patients
* Pregnant patients
* Pelvic organ prolapse stage greater than 2
* Patients with immunosuppression due to underlying medical conditions
* Recent antibiotic treatment within one week of the procedure

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 138 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Risk of post operative urinary tract infections (UTI) | 6 weeks after the procedure
  Intervention (pre-operative oral antibiotics) and placebo groups will be compared for the risk of post-operative UTIs following urethral bulking procedures performed in the operating room.
  Patients who have symptoms, concerning for UTI during the immediate 6 week postoperative period will be asked to give a urine sample for culture. UTIs which are culture proven and symptomatic will be treated per individual provider preference. Positive urine cultures will be defined as cultures with greater than 50,000 CFU for voided specimens and greater than 5,000 CFU for catheter specimens. If a patient's urine culture is positive for mixed flora and cannot be speciated further by our microbiology laboratory, they will be asked to present for a straight catheter specimen in the office for definitive diagnosis; this is an established protocol which is already standard in our practice. All positive cultures during this time period will be recorded.

SECONDARY OUTCOMES:
Drug Use and Side Effects | 6 weeks and 1 year after the procedure, up to 1 year
  Assessing if factors such as patient discharge with Intermittent self-catheterization (ISC)/indwelling foley or number of Bulkamid injection sites is correlated to improvement in SUI at 6 weeks and 1 year postoperatively.
Effects on higher patient satisfaction | 6 weeks and 1 year after the procedure, up to 1 year
  If any patient characteristics are associated with higher patient satisfaction following the procedure.
  Following the procedure, patients will be asked to complete a survey compromising of the Pelvic Floor Disability Index/Urinary Distress Inventory - Short Form (PFDI/UDI-6), the MESA questionnaire and an extended Visual Analogue Scale (VAS; scale of 0 or extremely unsatisfied to 100 or extremely satisfied). Patients will be given a paper copy of the survey at their 6 week post-operative appointment as well as an online link to complete the survey. This same survey will then be administered again approximately 1 year after the patient's procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Taege, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Female Pelvic Medicine and Reconstructive Surgery, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No